CLINICAL TRIAL: NCT03663023
Title: Band Adhesions in Relation to Previous Abdominal Surgery - a Retrospective Analysis of Risk Factors
Brief Title: Band Adhesions in Relation to Previous Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: Adhesions2018vgr
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Surgical Adhesions; Intestinal Obstruction; Surgery Induced Tissue Adhesions
MeSH Terms: conditions — Tissue Adhesions; Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intestinal obstruction

SUMMARY:
This study investigates the prevalence of previous abdominal surgery in a cohort of patients operated for bowel obstruction and analyzes the causes of obstruction discovered at surgery.

DETAILED DESCRIPTION:
Postoperative intra-abdominal adhesions are a common cause of small bowel obstruction. The extent of adhesions has been assigned to the magnitude of previous surgery. In a county hospital, with a catchment population of 120 000 inhabitants, records of operations performed for bowel obstruction over a period of 70 months were retrieved. Codes for bowel obstruction according to an International Classification of Diseases (ICD-10) will include: Intestinal adhesion with obstruction, Other and unspecified intestinal obstruction, Intestinal obstruction and Peritoneal adhesions. Amount of adhesions will be calculated in relation to previous surgery.

ELIGIBILITY:
Inclusion Criteria:

Subjects operated for bowel obstruction -from January 1st 2006 to October 31st 2011

Surgical codes for bowel obstruction:

* Intestinal adhesion with obstruction
* Other and unspecified intestinal obstruction
* Intestinal obstruction
* Unspecified and Peritoneal adhesions

Surgical procedures identified for bowel obstruction:

* Division of band adhesion
* Adhesiolysis
* Other separation of adhesion during bowel obstruction
* Laparotomy and reposition or detorsion of intestine.

Exclusion Criterias:

-Extra-peritoneal surgery such as inguinal or ventral hernia repair was excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: According to the protocol, 213 surgical procedures were identified. 17 procedures were excluded due to no bowel obstruction at surgery. Intestinal obstruction was evident in 196 procedures. These procedures were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2011-10-31 (Actual); Study Completion 2011-10-31 (Actual)

PRIMARY OUTCOMES:
Cause of bowel obstruction | 70 months
  Bowel obstruction; caused by adhesions, malignant disease, inflammation or other causes

IPD SHARING:
Plan to Share IPD: No